CLINICAL TRIAL: NCT02444611
Title: A Randomised, Controlled Trial Investigating the Influence of BCG (Bacillus Calmette-Guérin) and Hepatitis B Immunisation at Birth on Neonatal Immune Responses
Brief Title: A Trial Investigating the Influence of BCG and Hepatitis B Immunisation at Birth on Neonatal Immune Responses: The Early Life Vaccines and Immunity Study
Acronym: ELVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Royal Children's Hospital (Other); Mercy Hospital for Women, Australia (Other)
Responsible Party: Principal Investigator, Prof Nigel Curtis, Professor, Murdoch Childrens Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VAC/01 ELVIS
Record Dates: First submitted 2015-04-06; First posted 2015-05-14 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Innate Immune Response
Keywords: neonates; BCG; Hepatitis B vaccine; vaccines; immunity; immune response; Bacille- Calmette-Guerin
MeSH Terms: conditions — Hepatitis B | interventions — BCG Vaccine; Hepatitis B Vaccines; HB-VAX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): BCG vaccine, 0,05ml intradermally at birth
  Interventions: Drug: BCG Vaccine
- Group 2 (Active Comparator): BCG vaccine, 0,05ml intradermally at birth Hepatitis B vaccine, 5 micrograms, intramuscularly at birth
  Interventions: Drug: BCG Vaccine; Drug: Hepatitis B Vaccine
- Group 3 (Active Comparator): Hepatitis B vaccine, 5 micrograms, intramuscularly at birth
  Interventions: Drug: Hepatitis B Vaccine
- Group 4 (No Intervention): No birth vaccines

INTERVENTIONS:
Drug: BCG Vaccine — intradermal vaccination
  Other Names: BCG vaccine- Denmark strain; BCG Denmark; Statens Serum institute BCG vaccine; Mycobacterium bovis BCG vaccine, Danish strain, 1331; Bacillus-Calmette-Guerin
  Arms: Group 1; Group 2
Drug: Hepatitis B Vaccine — intramuscular vaccination
  Other Names: HB-Vax-II
  Arms: Group 2; Group 3

SUMMARY:
Neonatal morbidity and mortality from infectious diseases is of global concern. Childhood disease-specific immunisation is irrefutably linked to the decline in deaths from these targeted infections over the last century. However, neonatal immunisation is limited, in part, by the impaired adaptive immune function in this age group.

There is now an expanding body of evidence for heterologous ('non-specific') effects of various vaccines used in childhood. This refers to the immunomodulatory capabilities of vaccines to influence immune outcomes beyond the vaccine's specific targeted disease. The underlying immunological mechanisms responsible for these effects are incompletely understood, but evidence is mounting that the innate immune system is central to these observed effects.

This study is a randomised controlled trial designed to determine the influence of two commonly administered neonatal immunisations, BCG and Hepatitis B vaccine, given at birth, on the neonatal immune responses to non-specific antigens.

The investigators will recruit 200 newborns at the Mercy Hospital for Women in Melbourne, Australia over a 1-year period. These babies will be allocated randomly to one of 4 groups, receiving these 2 vaccines in different combinations, at 2 set time points. (at birth and 1 week post randomisation) A blood sample will be taken at 1-week post randomisation for in vitro immunological analyses.

This study will improve current understanding of the influence of vaccines on neonatal immunity and will help develop strategies exploiting beneficial heterologous ('non-specific') effects to improve protection against infection in the very young.

ELIGIBILITY:
Inclusion Criteria:

* English speaking parent
* Planned travel to a TB (Tuberculosis) endemic country within the infant's first 5 years of life
* An informed consent form must be signed and dated by the infant's mother after the nature of the study has been explained and prior to any study assessments/procedures
* The infant's mother has screened negative for HIV during this pregnancy
* The infant's mother has screened negative for Hepatitis B during this pregnancy
* There is no known household contact infected with Hepatitis B
* Born no earlier than eight weeks before estimated date of delivery
* Birth weight >1500g
* Delivered vaginally
* Singleton pregnancy

Exclusion Criteria:

* Known or suspected HIV infection
* Treatment with corticosteroids or other immunosuppressive therapy, including monoclonal antibodies against tumour necrosis factor---alpha (TNF---alpha) (e.g. infliximab, etanercept, adalimumab).
* Born to a mother treated with bDMARDs (biological Disease- Modifying Anti-Rheumatic drugs) (e.g. TNF---alpha blocking monoclonal antibodies) in the 3rd trimester
* Congenital cellular immunodeficiencies including specific deficiencies of the interferon gamma pathway
* Malignancies involving bone marrow or lymphoid systems
* Serious underlying illness including severe malnutrition
* Medically unstable
* Generalised septic skin disease and skin conditions such as eczema, dermatitis and psoriasis
* Significant febrile illness

Also excluded are infants with:

1. A mother who is immunosuppressed;
2. A mother who has received Intravenous immunoglobulins during her pregnancy
3. A family history of immunodeficiency;
4. Consanguineous parents.
5. Mother who is having a planned Caesarean Section
6. A home address more than 40 minutes drive from the Mercy hospital for Women and are unwilling to return to hospital for infant blood sampling

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cytokine concentrations (pg/ml) in response to in-vitro stimulation with a range of antigens | 7 (+-4) days post randomisation
  Four hours after blood samples are collected, they will be stimulated with different concentrations of infective antigens for 20hrs. (eg killed S.aureus, S. pneumoniae, E. Coli, Haemophilus Influenza B, Group B streptococcus, C. albicans), BCG, Hepatitis B sAg). Cytokine expression will be analysed in supernatants by Luminex -based multiplex assays.
  The cytokines that will be measured:
  Interleukin-1 beta, Interleukin-1ra, Interleukin-6, Interleukin-8, Macrophage/Monocyte Chemoattractant Protein-1(MCP-1), Macrophage Inflammatory Protein (MIP) -1 alpha, MIP-1 beta, Interferon(IFN) gamma, Interleukin-10, Macrophage migration inhibitory factor (MIF), Monokine induced by interferon (MIG), Tumour necrosis factor (TNF) alpha

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Curtis, MBBS,PHD, Principal Investigator — Royal Children's Hospital
Locations (1):
- Mercy Hospital for Women, Heidelberg, Victoria, Australia